CLINICAL TRIAL: NCT04575090
Title: 7 Tesla MRI Study in Patients With Statin Related Muscle Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Garg, Abhimanya, M.D. (Individual); Prishant Mishra (Unknown); Jimin Ren (Unknown)
Responsible Party: Principal Investigator, Zahid Ahmad, Associate Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 012016-017
Record Dates: First submitted 2020-05-15; First posted 2020-10-05 (Actual); Results first posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-04

CONDITIONS: Statin-related Muscle Pain; Muscle Aches; Muscle Weakness; Muscle Cramp; Muscle Stiffness
MeSH Terms: conditions — Myalgia; Muscle Weakness; Muscle Cramp | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Observational Arm) (No Intervention): Patients in substudy 1 will be identified by the PI from the clinic as individuals who are currently experiencing statin related muscle complaints or who have had severe reactions to statins in the past. There is going to be only one visit which will last for apprximately 3.5 hrs. Subjects will have height, weight and vitals measured. They will be asked pain and and demographic questionnaire. They will have their blood draw and will undergo MRS.
- Arm 2 (Interventional Experimental Arm) (Experimental): Subjects with statin related muscle complaints were enrolled in this arm and will have 3 visits. First visit is screening visit which will last for about 2 hrs and the next 2 visits will last for about 3.5 hrs. The screening visit will occur 2 weeks prior to visit 1.
  Subjects will have height, weight and vitals measured. They will be asked pain and and demographic questionnaire. They will have their blood draw and will undergo MRS.
  Some volunteers who do/do not regularly exercise or are/are not active in sports may be asked to exercise prior to the MRS. This exercise may be in the form of hand grasps, toe-raises, bicycling on a stationary bike or walking on a treadmill. Exercise will be limited to up to one hour, during which time the subject's vital signs and blood oxygenation will be monitored. During the scan, the subject's heart rate and respiratory rate may be monitored
  Interventions: Drug: Simvastatin
- Arm 3 (Interventional Control Arm) (Experimental): Subjects with no statin related muscle complaints were enrolled in this arm and will have 3 visits. First visit is screening visit which will last for about 2 hrs and the next 2 visits will last for about 3.5 hrs. The screening visit will occur 2 weeks prior to visit 1.
  Subjects will have height, weight and vitals measured. They will be asked pain and and demographic questionnaire. They will have their blood draw and will undergo MRS.
  Some volunteers who do/do not regularly exercise or are/are not active in sports may be asked to exercise prior to the MRS. This exercise may be in the form of hand grasps, toe-raises, bicycling on a stationary bike or walking on a treadmill. Exercise will be limited to up to one hour, during which time the subject's vital signs and blood oxygenation will be monitored. During the scan, the subject's heart rate and respiratory rate may be monitored
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40 mg daily.
  Arms: Arm 2 (Interventional Experimental Arm); Arm 3 (Interventional Control Arm)

SUMMARY:
Roughly 5-10% of statin-treated patients report muscle pain, aches, weakness, cramps, stiffness, or "heaviness" - typically occurring symmetrically in the legs. For healthcare providers, the major diagnostic challenge is to unambiguously link these symptoms to statin use, especially since some patients can have normal serum creatine kinase (CK) levels despite demonstrable weakness and muscle biopsy proven statin-induced myopathy .

No well accepted, standardized, or Food and Drug Administration (FDA)-endorsed diagnostic method exists for statin-induced muscle injury. This lack of an objective diagnostic methodology blocks vertical advancement of the field.

The successful completion of this project will develop in vivo techniques that will provide insight into how statins affect muscle metabolism and help establish a methodology to objectively diagnose muscle injury due to statins. The development of an MRS technique will allow for in-vivo analyses and the data accumulated here will serve as preliminary data for futher extramural funding of studies with much larger sample sizes. Ultimately, this focus of research will lead to improved diagnosis and treatment of patients with statin-related muscle complaints, which is central to obtaining the cardiovascular risk reduction from lipid-lowering drugs.

DETAILED DESCRIPTION:
The goal of the first study will be to generate hypothesis regarding the long-term effects of statin in muscles by studying 7T MRS findings in patients who are currently experiencing statin-related muscle complaints or who have a history of severe reactions to statins (i.e. rhabdomyolysis, anti-HMGCR-associated autoimmune myopathy, or CK elevation > 10 times the upper limit of normal). We anticipate enrolling roughly 5 such patients. The protocol involves a single visit for a blood draw and MRS of calf muscle. The data will be compared to historical controls provided by the Advanced Imaging Research Center.

Second, we will study the effect of short-term statin administration in 5 patients with a history of statin related muscle complaints and 5 controls with no statin related muscle complaints . Controls will be matched for age, weight, and body mass index. Patients will undergo a wash-out of lipid lowering drugs followed by a challenge with simvastatin 40 mg daily (similar to a statin withdrawal and rechallenge). We chose simvastatin since it is the most common statin that caused myopathy according to our preliminary data (as well as most other published reports). Each patient will have 5 visits. The screening visit will involve a review of inclusion/exclusion criteria, blood draw, questionnaire, and instructions to withhold all lipid lowering drugs until visit 1. Any patient with known antibodies to HMGCR will be excluded from the remainder of the study.

Visit 1 will occur 2 weeks after stopping all lipid lowering drugs. A minimum 2 week period off lipid lowering drugs is required to allow clearance of any medication from the systemic circulation. Patients will undergo MRS of the calf muscle and a blood draw. Patients will then start simvastatin 40 mg daily.

ELIGIBILITY:
Inclusion Criteria:

Adults age >18 yrs or <80 yrs Patients reporting complaints of statin-associated muscle symptoms, aches, weakness, cramps, or stiffness of legs.

Exclusion Criteria:

Patients who drink large quantities of grapefruit juice (>1 quart daily)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03-05 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2021-06-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Arm 1 is an observational study. No intervention involved. No data was collected for arm 1
Groups:
- No Intervention: Arm 1 (Observational Arm): Patients in Arm 1 will be identified by the PI from the clinic as individuals who are currently experiencing statin related muscle complaints or who have had severe reactions to statins in the past. There is going to be only one visit which will last for apprximately 3.5 hrs. Subjects will have height, weight and vitals measured. They will be asked pain and and demographic questionnaire. They will have their blood draw and will undergo MRS.
- Experimental: Arm 2 (Interventional Experimental Arm): Subjects with statin related muscle complaints were enrolled in this arm and will have 3 visits. First visit is screening visit which will last for about 2 hrs and the next 2 visits will last for about 3.5 hrs. The screening visit will occur 2 weeks prior to visit 1.
  Subjects will have height, weight and vitals measured. They will be asked pain and and demographic questionnaire. They will have their blood draw and will undergo MRS.
  Some volunteers who do/do not regularly exercise or are/are not active in sports may be asked to exercise prior to the MRS. This exercise may be in the form of hand grasps, toe-raises, bicycling on a stationary bike or walking on a treadmill. Exercise will be limited to up to one hour, during which time the subject's vital signs and blood oxygenation will be monitored. During the scan, the subject's heart rate and respiratory rate may be monitored
- Experimental: Arm 3 (Interventional Control Arm): Subjects with no statin related muscle complaints were enrolled in this arm and will have 3 visits. First visit is screening visit which will last for about 2 hrs and the next 2 visits will last for about 3.5 hrs. The screening visit will occur 2 weeks prior to visit 1.
  Subjects will have height, weight and vitals measured. They will be asked pain and and demographic questionnaire. They will have their blood draw and will undergo MRS.
  Some volunteers who do/do not regularly exercise or are/are not active in sports may be asked to exercise prior to the MRS. This exercise may be in the form of hand grasps, toe-raises, bicycling on a stationary bike or walking on a treadmill. Exercise will be limited to up to one hour, during which time the subject's vital signs and blood oxygenation will be monitored. During the scan, the subject's heart rate and respiratory rate may be monitored
Period: Overall Study
Arm/Group | No Intervention: Arm 1 (Observational Arm) | Experimental: Arm 2 (Interventional Experimental Arm) | Experimental: Arm 3 (Interventional Control Arm)
Started | 0 | 7 | 1
Completed | 0 | 5 | 1
Not Completed | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Arm 1 is an observational study. No intervention involved. No data was collected for arm 1
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention: Arm 1 (Observational Arm) | Experimental: Arm 2 (Interventional Experimental Arm) | Experimental: Arm 3 (Interventional Control Arm) | Total
Number analyzed (Participants) | 0 | 7 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 1 | 3
  >=65 years | 0 | 5 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 0 | 4
  Male | 0 | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 0 | 2 | 0 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Median (Standard Deviation); unit: kg/m^2] |  | 31.2 (6.0) | 22 (0) | 26.6 (6)
Phospho Creatnine/ Adenosine Triphosphate (PCr/gATP) [Mean (Standard Deviation); unit: ratio] — The PCr/gATP represents the ratio of 31P MRS signal intensity between phosphocreatine (PCr) and ATP ("gATP" means ATP phosphate at gamma position). The PCr/ATP ratio is an index of immediate energy reserve in the skeletal muscle. The higher the PCr/ATP ratio, the more the energy reserve the skeletal muscle has for handling immediate energy demand, so that ATP will not be exhausted. In other words, PCr is coupled to ATP (through creatine kinase) to maintain energy homeostasis in skeletal muscle and other high energy demanding tissues (brain and heart). Population: Arm 2 : Data of 5 subjects were analyzed. For the remaining 2 - data was not analyzable.
  ratio |  | 4.765 (0.459) | 4.344 (0) | 12.85 (0.29)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pre- and Post-phosphocreatine Relaxation Time
Description: Measure differences in pre- and post-phosphocreatine relaxation time in SAMS (Statin Associated Muscle Symptoms) patients on simvastatin compared to placebo.
Time Frame: Baseline, 10 Weeks
Population: Arm 1 is an observational study. No intervention involved. No data was collected for arm 1 Arm 2: Data of 5 subjects were analyzed. For the remaining 2 - data was not analyzable.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- No Intervention: Arm 1 (Observational Arm): Patients in arm 1 will be identified by the PI from the clinic as individuals who are currently experiencing statin related muscle complaints or who have had severe reactions to statins in the past. There is going to be only one visit which will last for apprximately 3.5 hrs. Subjects will have height, weight and vitals measured. They will be asked pain and and demographic questionnaire. They will have their blood draw and will undergo MRS.
  Some volunteers who do/do not regularly exercise or are/are not active in sports may be asked to exercise prior to the MRS. This exercise may be in the form of hand grasps, toe-raises, bicycling on a stationary bike or walking on a treadmill. Exercise will be limited to up to one hour, during which time the subject's vital signs and blood oxygenation will be monitored. During the scan, the subject's heart rate and respiratory rate may be monitored
Arm/Group | No Intervention: Arm 1 (Observational Arm) | Experimental: Arm 2 (Interventional Experimental Arm) | Experimental: Arm 3 (Interventional Control Arm)
Number analyzed (Participants) | 0 | 5 | 1
milliseconds |  | 5.58 (1.6) | 5.083 (0)

ADVERSE EVENTS:
Time Frame: Data was collected over a period of 6 months.
Description: Arm 1 is an observational study. No intervention involved. AEs were not assessed in this arm 1.
Arm/Group | No Intervention: Arm 1 (Observational Arm) | Experimental: Arm 2 (Interventional Experimental Arm) | Experimental: Arm 3 (Interventional Control Arm)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/7 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/7 | 0/1

LIMITATIONS AND CAVEATS:
There was an error / typo in the explanation that was provided at the time of the previous submission within this section.

Hence to clarify and confirm - Arm 1 is an observational study. No intervention is involved. No data was collected for arm 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT04575090/Prot_SAP_000.pdf